CLINICAL TRIAL: NCT06690307
Title: The Efficacy and Safety of Oxycodone in Patient-controlled Intravenous Analgesia After Laparoscopic Hysterectomy
Brief Title: Oxycodone Versus Sufentanil in Patient-controlled Intravenous Analgesia After Laparoscopic Hysterectomy
Acronym: Oxycodone
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Principal Investigator, Siyuan Liu, Principal Investigator, Affiliated Hospital of Nantong University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-K115-01
Record Dates: First submitted 2024-11-09; First posted 2024-11-15 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Laparoscopic Hysterectomy
Keywords: oxycodone; patient-controlled intravenous analgesia; laparoscopic hysterectomy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sulfentanil group (Active Comparator): Participants in the active comparator group will receive sulfentanil for PCIA.
  Interventions: Procedure: patient controlled intravenous analgesia(PCIA)
- oxycodone group (Experimental): Participants in the experimental group will receive oxycodone for PCIA.
  Interventions: Procedure: patient controlled intravenous analgesia(PCIA)

INTERVENTIONS:
Procedure: patient controlled intravenous analgesia(PCIA) — Patients will receive sulfentanil for PCIA.
  Arms: sulfentanil group
Procedure: patient controlled intravenous analgesia(PCIA) — Patients will receive oxycodone for PCIA.
  Arms: oxycodone group

SUMMARY:
This study is designed to evaluate the efficacy and safety of hydrocodone in patient-controlled intravenous analgesia (PCIA) during gynecological laparoscopy, thus to explore suitable PCIA scheme to optimize postoperative pain management for patients undergoing gynecological laparoscopic surgeries.

DETAILED DESCRIPTION:
The controlled group will receive sulfentanil for PCIA, and the test group will receive hydrocodone for PCIA. NRS scores at 1, 6, 24 and 48 hours post-surgery will be recorded. The usage of rescue analgesics and adverse events will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* selective laparoscopic hysterectomy
* general anesthesia
* ASA classification I - III
* aged 18 - 65 years

Exclusion Criteria:

* allergy to oxycodone or any other drugs will be used in the study
* preoperative opioids medication
* opioids abuse
* hepatic or renal dysfunction
* cardiovascular or pulmonary dysfunction
* lack of full civil capacity or refuse to participate

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
NRS scores | 6 hours after surgery
  Postoperative pain will be evaluated on a 11point number rating scale (NRS): 0 means no pain; and 10 means worst pain imaginable.

SECONDARY OUTCOMES:
NRS scores | 1, 24, 48 hours after surgery
  Postoperative pain will be evaluated on a 11point number rating scale (NRS): 0 means no pain; and 10 means worst pain imaginable.
rescue analgesics usage | from the end of surgery to the first usage (up to 48 hours post-surgery)
  time to the first use of rescue analgesics
PCIA pressing times | 48 hours after surgery
  total pressing times and effective pressing times
anal exhaust time | from the end of surgery to the first anal exhaust (up to 48 hours post-surgery)
adverse events | within 48 hours after surgery
  dizziness, drowsiness, nausea and vomiting, intestinal paralysis, skin itching, respiratory depression, intestinal obstruction, severe allergic reactions, and serious cardiovascular adverse events
NRS scores | 30 days after surgery
  Postoperative pain will be evaluated on a 11point number rating scale (NRS): 0 means no pain; and 10 means worst pain imaginable.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided